CLINICAL TRIAL: NCT05907317
Title: Safeguarding the Brain of Our Smallest Children-IIIv (SafeBoosC-IIIv): Cerebral Oximetry Versus Usual Care in Mechanically Ventilated Newborns
Brief Title: Safeguarding the Brain of Our Smallest Children-IIIv (SafeBoosC-IIIv)
Acronym: SafeBoosC-IIIv
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SafeBoosC-IIIv
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Hypoxia; Infant, Newborn, Diseases
Keywords: Near-infrared spectroscopy; Randomised clinical trial; Mechanical ventilation
MeSH Terms: conditions — Hypoxia; Infant, Newborn, Diseases

STUDY DESIGN:
Intervention Model Description: The trial will recruit 1610 babies in step one. Randomisation will continue until 3000 babies are recruited in step two.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Step one: The primary outcome will be assessed by a blinded investigator. The principal investigator from each centre must develop a local blinding procedure, describing how blinding is achieved. To support the principal investigators in this work, a Standard Operation Procedure with suggestions for blinding procedures will be developed. Data managers, statisticians, and conclusion drawers will be blinded.
  Step two: Due to the nature of the experimental intervention, clinical staff and the parents will not be blinded to group allocation. Thus, the primary outcome will not be blinded in cases when it relies on parental reporting. If there is no contact with the parents, or if they do not return the questionnaire, data will be collected from health care records. Investigators reviewing the health care records will, if possible, be blinded to the allocated intervention. Data managers, statisticians, and conclusion drawers will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebral oximetry + usual care (Experimental)
  Interventions: Device: Cerebral oximetry monitoring device; Other: Usual care
- Usual care (Other): The control group will receive mechanical ventilation without access to cerebral oximetry and the SafeBoosC treatment guideline. If the newborn is cared for outside the neonatal unit at any time, e.g. during surgery, cerebral oximetry may or may not be used, as decided by the responsible physician there
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Cerebral oximetry monitoring device — Participants in the experimental group will be monitored with cerebral oximetry, if possible before or, as soon as possible and within six hours after initiation of invasive mechanical ventilation. Cerebral oximetry will be continued until 1) the cardio-pulmonary function has been stabilised as indicated by the need for respiratory and circulatory support and evaluated by the responsible physician, 2) extubation, 3) until 28 days after birth, or 4) until death. Randomisation will only direct the use of cerebral oximetry during the first invasive mechanical ventilation episode. Cerebral oximetry will be used to minimise cerebral hypoxia by modifying clinical care according to the SafeBoosC treatment guideline and monitoring as usual.
  Arms: Cerebral oximetry + usual care
Other: Usual care — Treatment as usual

SUMMARY:
The objective of the SafeBoosC-IIIv trial is to assess benefits and harms of cerebral oximetry in newborns receiving invasive mechanical ventilation. The hypothesis is that:

i. Cerebral oximetry added to usual care versus usual care alone in newborns receiving invasive mechanical ventilation will increase the number of hospital-free days within 90 days of randomisation.

ii. The intervention will decrease a composite outcome of death or moderate to severe neurodevelopmental disability and/or increase the mean PARCA-R non-verbal cognitive score at two years of corrected age.

DETAILED DESCRIPTION:
SafeBoosC-IIIv will be an investigator-initiated, multinational, randomised, pragmatic phase III clinical trial. The trial will be conducted in two steps. In step one, 1,610 newborns will be randomised, and the outcomes will be assessed 90 days after randomisation. Funding has been obtained for step one. If further funding is obtained, we will continue to include newborns until a total of 3,000 newborns are randomised and then follow them up at two years of corrected age (step two).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age more than or equal to 28+0
* Postnatal age less than 28 days
* Expected to receive invasive mechanical ventilation (intubation) for at least 24 hours, as judged by the physician intending to randomise
* Parental informed consent unless the centre has chosen to use 'opt-out' or deferred consent as consent method
* A cerebral oximeter available so monitoring can be started within six hours after initiation of invasive mechanical ventilation

Exclusion Criteria:

* Suspicion of or confirmed brain injury or disorder (e.g. severe hypoxic-ischemic encephalopathy, intraventricular haemorrhage grade 3 or 4, cerebral malformation, genetic or metabolic disease)
* Suspicion or diagnosis of congenital heart malformations likely to require surgery

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1610 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Hospital-free days within 90 days of randomisation | 90 days
  Primary outcome for step one
A composite of death from any cause or moderate to severe neurodevelopmental disability | 2 years
  Co-primary outcome for step two
  A composite of death from any cause or moderate to severe neurodevelopmental disability at two years of corrected age. Moderate to severe neurodevelopmental disability will be defined as one or more of the following
  1. cerebral palsy with Global Motor Function Classification System level 2 or higher;
  2. a Parent Report of Children's Abilities-Revised (PARCA-R) non-verbal cognitive function score (range 0-34, higher score means better outcome) below -2 standard deviations (SD);
  3. hearing loss corrected with aids or worse; or
  4. vision impairment defined as moderately reduced vision of one eye, or only being able to perceive light or light reflecting objects; or blind in one eye with good vision in the contralateral eye.
Parental questionnaires | 18-30 months
  Co-primary outcome for step two: Parental questionnaires completed between 18-30 months' corrected age as well as available data from at least 12 months' corrected age from health care records, including standardised neurodevelopmental assessments, will be used to assess mortality and neurodevelopment.
  • Non-verbal cognitive score of Parent Report of Children's Abilities-Revised (PARCA-R), a parental questionnaire, at two years of corrected age (range 0-34, higher score means better outcome).

SECONDARY OUTCOMES:
Proportion of participants with a serious adverse event | 90 days
  Secondary outcome for step one: Proportion of participants with one or more Serious Adverse Events within the 90 days of randomization, i.e. one or more of the following:
  Death from any cause Bronchopulmonary dysplasia (BPD) Any brain injury diagnosed by imaging Seizures treated with antiepileptic medicine Haemodynamic insufficiency that needs cardiovascular support Spontaneous bowel perforation or necrotising enterocolitis (NEC) Bells grade 2 or more Nosocomial infection Extra Corporal Membrane Oxygenation (ECMO) Renal replacement therapy
Invasive mechanical ventilation-free days within 90 days of randomisation | 90 days
  Secondary outcome for step one

OTHER OUTCOMES:
Late onset sepsis | 90 days
  Exploratory outcome for step one
Invasive mechanical ventilation-related infection | 90 days
  Exploratory outcome for step one
Cerebral palsy | 2 years
  Exploratory outcome for step two: defined as Global Motor Function Classification System level 2 or above, at two years of corrected age.
Sensory deficit | 2 years
  exploratory outcome for step two: defined as any degree of vision or hearing impairment, at two years of corrected age.
All-cause mortality | 2 years
  Exploratory outcome for step two: Mortality at two years of corrected age.
Use of daily medication | 2 years
  Exploratory outcome for step two: Use of medication during the last two months, at two years of corrected age.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vestager ML, Hansen ML, Rasmussen MI, Hahn GH, Hyttel-Sorensen S, Pellicer A, Heuchan AM, Hagmann C, Dempsey E, Dimitriou G, Pichler G, Naulaers G, Fuchs H, Tkaczyk J, Mintzer J, Fumagalli M, Nesargi S, Fredly S, Szczapa T, Gluud C, Jakobsen JC, Greisen G. The effects of cerebral oximetry in mechanically ventilated newborns: a protocol for the SafeBoosC-IIIv randomised clinical trial. Trials. 2023 Oct 28;24(1):696. doi: 10.1186/s13063-023-07699-x. PMID 37898759
- [Derived] Petersen JJ, Kamp CB, Olsen MH, Hansen ML, Thorlund K, Pellicer A, Naulaers G, Dempsey E, Hahn GH, Andersen PB, Rasmussen MIS, Pichler G, Dimitriou G, Szczapa T, Ognean ML, Nesargi S, Musante G, Chalak L, Di Maio M, Lakhwani J, Procianoy RS, Tkaczyk J, Fuchs H, Cetinkaya M, Hagmann C, Popat H, Fabres J, Wang L, Schmolzer G, Piris-Borregas S, Mohora R, Zafra P, Sarafidis K, Alsina-Casanova M, Baik-Schneditz N, Lopez LS, Griesmaier E, Hatzidaki E, Shashidhar A, Dassios T, Arruza L, Greisen G, Jakobsen JC. Treatment guided by cerebral oximetry in mechanically ventilated newborns: a statistical analysis plan for step one of the SafeBoosC-IIIv randomised clinical trial. Trials. 2025 Dec 18. doi: 10.1186/s13063-025-09387-4. Online ahead of print. PMID 41413912
- See also: Official website of the trial — https://safeboosc.eu
- Available data/document: Study Protocol — https://www.rigshospitalet.dk/english/departments/juliane-marie-centre/department-of-neonatology/research/safeboosc-iiiv/Pages/protocol.aspx